CLINICAL TRIAL: NCT04298294
Title: The Effect of Using of Injectable Platelet Rich Fibrin on Filling the Gap of Immediate Dental Implant in the Esthetic Zone
Brief Title: Using of Injectable Platelet Rich Fibrin on Filling the Gap of Immediate Dental Implant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Bassant Mohye, Principal Investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Bassant Mohye
Record Dates: First submitted 2020-02-29; First posted 2020-03-06 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Bone Loss
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Intervention Model Description: Group I (study group)8 patients undergo flapless single immediate implant placement surgery with filling the gap distance with i-PRF& bone graft
  Group II (control group) 8 patients undergo flapless single immediate implant placement surgery with filling the gap distance with bone graft
Who Masked: Investigator, Outcomes Assessor
Masking Description: double blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- injectable platelet rich fibrin group (Experimental): 8 patients undergo flapless single immediate implant placement surgery with filling the gap distance with i-PRF& bone graft
  Interventions: Other: injectable platelet rich fibrin
- no injectable platelet rich fibrin group (No Intervention): 8 patients undergo flapless single immediate implant placement surgery with filling the gap distance with bone graft

INTERVENTIONS:
Other: injectable platelet rich fibrin — biologic activator
  Arms: injectable platelet rich fibrin group

SUMMARY:
The effect of using of i-PRF (injectable platelet rich fibrin) on filling the gap of immediate dental implant in the esthetic zone

DETAILED DESCRIPTION:
Grouping the samples: (sixteen patients was recruited from the outpatient clinic of Oral Medicine, Periodontology, Diagnosis and Radiology Department, Faculty of Dentistry, Ain Shams University).

The sixteen patients assigned to group 1 or group 2 will be randomly allocated using flip of a coin into one of the 2 treatment modalities.

Primary objective:

Radiograhic evaluation of the effect of i-PRF on filling the buccal gap distance between the immediately placed dental implant and the surrounding bone.

Secondary objective:

Esthetic evaluation of the effect of i-PRF on the soft tissue around immediately placed dental implant.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult patient.
* Age from 20-50 years old
* Patients must be free of any systemic disease which could influence the surgical procedure.
* Tooth involved in the esthetic zone.
* Sufficient hard and soft tissue volume in vertical and buccolingual 6. Natural teeth adjacent to the involved tooth were required to be free from infection.
* Controlled oral hygiene.
* Indication for tooth extraction included;

  * Endodontic failures
  * Untreatable caries> Non- restorable teeth
  * Vertical root fracture
  * Remaining roots
* The decision to proceed with the implant placement was made after tooth extraction and probing of the extraction socket which revealed:

  * The presence of intact facial bone.
  * Compliance with all requirements in the study and signing the informed consent.

Exclusion Criteria:

* Patient had surgeries in the same site during the last 6 months prior to the surgery.
* Severe vertical bone loss (socket type lll or type lV).
* Presence of acute dento-alveolar infection or periodontal affected of involved tooth.
* Pregnant and lactating females.
* Smokers.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2018-02-16 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Radiograhic evaluation of the effect of i-PRF on filling the buccal gap distance between the immediately placed dental implant and the surrounding bone. | 6 months follow up
  density, vertical and horizontal assessment of labial plate
Radiographic analysis | 6 months follow up
  vertical assessment of labial plate
Radiographic analysis | 6 months follow up
  density of labial plate

SECONDARY OUTCOMES:
Esthetic evaluation of the effect of i-PRF on the soft tissue around immediately placed dental implant | 6 months follow up
  pink esthetic score

CONTACTS AND LOCATIONS:
Locations (1):
- Bassant Mohye, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No